CLINICAL TRIAL: NCT06351904
Title: A Phase Ⅰ, Open Label, Multi-center Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of RAG-01 in Patients With Non-muscle-invasive Bladder Cancer (NMIBC) Who Have Failed Bacillus Calmette Guérin (BCG) Therapy
Brief Title: A Study of RAG-01 in Patients With Non-muscle-invasive Bladder Cancer (NMIBC) Who Have Failed Bacillus Calmette Guérin (BCG) Therapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ractigen Therapeutics. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RAG-01-01
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Non-Muscle-Invasive Bladder Cancer (NMIBC)
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- RAG-01 dose escalation and dose expansion (Experimental): The starting dose of RAG-01 is 30mg, and there are 4 dose cohorts, including 30mg, 100mg, 300mg, 600mg, respectively. Each eligible subject will be distributed into one cohort. Safety and pharmacokinetics are assessed at each dose level.
  Interventions: Drug: RAG-01

INTERVENTIONS:
Drug: RAG-01 — RAG-01 is a therapeutic small activating RNA (saRNA) duplex molecule comprised of two partially chemically modified complementary oligonucleotide strands.

SUMMARY:
This is an open label, multi-center study to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary efficacy of RAG-01 in patients with NMIBC who have failed BCG therapy.

DETAILED DESCRIPTION:
This study includes a dose escalation and a dose expansion. The dose escalation part will adopt a '3+3' dose escalation design. Additional subjects may be enrolled to have approximately 12 patients in each selected dose level for RDE determination. A randomized, open label, parallel-arm study will be conducted during the dose expansion part for further dose exploration. Approximately 40-60 subjects will be randomized in a 1:1 ratio into two treatment groups with dose levels selected from dose escalation part of the study. Randomization will be stratified based on disease type at enrollment (papillary-only vs. CIS). A dose selection analysis will be performed to assess safety, efficacy, PK, and PD, where applicable, to determine the optimal dose for RAG-01. The main study period includes the screening, initial treatment and DLT assessment period, second and third treatment period and the sequential follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the study and have signed the informed consent form;
2. Any adult ≥ 18 years old;
3. Pathologically confirmed high grade NMIBC defined as grade 2 or grade 3 disease;
4. Expected survival ≥ 6 months;
5. ECOG PS ≤2;
6. Sufficient organ functions, as defined below:

   Investigations Hematology Absolute Neutrophil Count (ANC): ≥ 1.5 x 109/L Hemoglobin: ≥ 90 g/L Platelet: ≥ 100 x 109/L Liver Function Serum bilirubin: ≤ 1.25×ULN or 2.5×ULN（with Gilbert syndrome） AST & ALT: ≤ 2.5×ULN Renal Function Creatinine Clearance (Cockcroft-Gault equation): ≥ 30 mL/min
7. Subject must be able to tolerate catheterization;
8. Female subject of childbearing potential and her spouse must use adopt effective contraception (non-pharmacological contraception required) from signing informed consent to within 6 months after the last instillation;

Exclusion Criteria:

1. Subject who is allergy to RAG-01 or similar products;
2. Except for TURBT, the subject received other anti-tumor treatments, and the last administration date is within ≤ 21 days or 5 half-lifes whichever is shorter from the date of signing ICF;
3. Subject with imaging examination diagnosed extravesical metastasis, including ureter and urethra;
4. Subject has other malignancies within the past 3 years, except for adequately treated carcinoma of the cervix, basal or squamous cell carcinomas of the skin, or adenocarcinoma of the prostate that has been surgically treated with a post-treatment PSA that is non-detectable;
5. The following illnesses have not been relieved to CTCAE 0-1:

   1. Uncontrolled acute and chronic infections, such as pneumonia, biliary tract infection, hepatitis B virus infection and hepatitis C virus infection;
   2. Dyspnea;
   3. Acute and chronic kidney injury, and inflammation;
   4. Urinary incontinence;
   5. Urinary frequency;
   6. Urinary tract obstruction (except benign prostatic hypertrophy);
6. Subject could not hold the urine for at least 90 mins due to any reason;
7. New York Heart Association (NYHA) 3 or 4 grade;
8. Coronary heart disease related symptoms have not been relieved to CTCAE 0-1, including: myocardial infarction, unstable angina pectoris, congestive heart failure and arrhythmia;
9. Subject with QTc >470 msec.
10. Cerebrovascular accidents have not been relieved to CTCAE 0-1;
11. HIV positive; Active hepatitis B or C. For active HBV, it's defined as HBsAg positive with HBV DNA ≥ ULN, for active HCV, it's defined as HCV antibody positive with HCV RNA ≥ ULN, respectively.
12. Subject is pregnant or lactating during the treatment period;
13. History of central nervous system or psychiatric disorders, e.g., epilepsy or dementia;
14. Other severe systemic diseases which might compromise the subject's compliance to the study, e.g., uncontrolled diabetes, gastrointestinal disorders, and renal diseases;
15. Any other situations which are judged by the investigator, would exposure the subject to unnecessary risk, therefore he/she is not eligible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2028-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of RAG-01 in patients with non-muscle-invasive bladder cancer (NMIBC) | From the screening to 6 months after the first instillation of RAG-01
  Adverse events (AEs), serious adverse events (SAEs), and adverse events during treatment (TEAEs)
Maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D) of RAG-01 | Within 21 days after first instillation
  Dose-limiting toxicity (DLT)

CONTACTS AND LOCATIONS:
Overall Officials: Laurence Krieger, MBCHB, Principal Investigator — GenesisCare, 7 Westbourne Street, St Leonards, NSW 2065, Australia
Locations (3):
- Australia (3):
  - GenesisCare North Shore, St Leonards, New South Wales
  - The Royal Melbourne Hospital, Melbourne, Victoria
  - Peninsula & South Eastern Haematology and Oncology Group, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No